CLINICAL TRIAL: NCT00306267
Title: A Pilot Study to Evaluate the Safety and Efficacy of PROCRIT (Epoetin Alfa) 80,000 Units Once Every Four Weeks (Q4W) vs. 40,000 Units Once Every Two Weeks (Q2W) in Cancer Subjects With Non-Chemotherapy Anemia (NCA)
Brief Title: A Study of PROCRIT (Epoetin Alfa) 80,000 Units (U) Once Every Four Weeks (Q4W) vs. 40,000 U Once Every Two Weeks (Q2W) in Cancer Patients Not Receiving Chemotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study stopped as it would not address important survival concerns raised in other recently conducted clinical studies.
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Ortho Biotech Products, L.P. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR010540
Record Dates: First submitted 2006-03-21; First posted 2006-03-23 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2010-03

CONDITIONS: Anemia; Cancer; Epoetin Alfa
Keywords: Anemia; non-chemotherapy-induced; non-radiation therapy-induced; cancer; non-myeloid
MeSH Terms: conditions — Anemia; Neoplasms | interventions — Epoetin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: epoetin alfa

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of PROCRIT (Epoetin alfa) administered by injection subcutaneously (SC, under the skin), at a dose of 80,000 U once every four weeks or 40,000 U once every two in anemic patients with cancer not receiving chemotherapy or radiation therapy.

DETAILED DESCRIPTION:
Epoetin alfa is an analogue (has the identical amino acid sequence) of erythropoetin, a hormone secreted by kidneys known to stimulate red blood cell production. Although epoetin alfa has been known to be effective in treatment of anemia associated with cancer chemotherapy, there are no specific formal guidelines on the use of epoetin alfa for the treatment of anemia in cancer patients not receiving chemotherapy or radiation therapy. Several prospective clinical trials investigating the efficacy of epoetin alfa in cancer-associated anemia included groups of patients not receiving chemotherapy where it was demonstrated that the use of epoetin alfa in this population was safe and effective in increasing hemoglobin (Hb) levels and reducing transfusion requirements. The optimal dosing regimen of epoetin alfa in cancer patients not receiving chemotherapy or radiation therapy remains unclear.

This 17-week study is a prospective, randomized, open-label, multi-center study to assess the safety and effectiveness of epoetin alfa in anemic patients with cancer not receiving chemotherapy or radiation therapy. Eligible patients with hemoglobin level <= 11 g/dL will receive epoetin alfa 40,000 U once every 2 weeks for 15 weeks or 80,000 U once every 4 weeks for 13 weeks. The study hypothesis are that there are no long-term safety concerns of epoetin alfa administered at these two dosing regimens and that both dosing regimens are equally effective in this patient population. Eligible patients with hemoglobin levels <= 11 g/dL will receive epoetin alfa 40,000 U once every 2 weeks for 15 weeks or 80,000 U once every 4 weeks for 13 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have "Active non-myeloid cancer malignancy" or incurable cancer with a life expectancy of 6 months or more
* Patients may also have had cancer treatment within the past 2 years but no chemotherapy or radiation therapy within the past 8 weeks prior to enrollment
* must be >= 18 years of age and must not be receiving or planning to receive cytotoxic chemotherapy or external beam radiotherapy during the study period
* must have a baseline Hb <= 11 g/dL.
* Patients with reproductive potential must be practicing an effective method of birth control and women cannot be pregnant or breast-feeding during the study period
* Patients must be able to comply with all requirements of the study (i.e. study visit schedules) and patients (or their legally authorized representatives) must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study

Exclusion Criteria:

* Patients receiving or planning to receive chemotherapy or radiation therapy within 8 weeks of study entry
* Anemia due to factors other than cancer
* Previous treatment with epoetin alfa or any form of erythropoietin during the previous 1 month or received an experimental drug or device within past 30 days
* Known hypersensitivity to mammalian-cell derived products or to human albumin
* Untreated known central nervous system (CNS) metastases
* Uncontrolled or clinically severe disease of the pulmonary, cardiovascular, endocrine, neurologic, gastrointestinal, or genitourinary systems not attributable to underlying malignancy or chemotherapy
* History of (within 12 months) deep venous thrombosis (DVT), pulmonary embolus (PE), or other venous thrombotic events, cerebrovascular accident (CVA), transient ischemic attack (TIA), Acute Coronary Syndrome (ACS) [unstable angina, myocardial infarction (MI)], or other arterial thrombosis
* Currently receiving therapeutic or prophylactic anticoagulants
* Transfusion of packed red blood cells within 28 days prior to the first dose of study drug, or planned stem cell harvest of bone marrow or high dose chemotherapy with stem cell transplant during study duration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2006-03; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint will be hematopoietic response, defined as >= 1 g/dL rise in hemoglobin from baseline.

SECONDARY OUTCOMES:
Secondary objectives are to assess the two dosing regimens on time-to-hematopoietic response and transfusion requirements. Safety assessments will include laboratory tests, blood pressure, physical examination and severity of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A Pilot Study to Evaluate the Safety and Efficacy of PROCRIT� (epoetin alfa) 80,000 Units Once Every 4 Weeks (q4w) vs. 40,000 Units Once Every 2 Weeks (q2w) in Cancer Subjects With Non-Chemotherapy Anemia (NCA) — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=716&filename=CR010540_CSR.pdf